CLINICAL TRIAL: NCT07211854
Title: Antithrombotic Strategies in Coronary Artery Dilatations and Aneurysms
Acronym: ASCADA
Status: Completed | Type: Observational
Sponsor: Franck Assayag (Other)
Responsible Party: Sponsor-Investigator, Franck Assayag, hospital practitioner, Versailles Hospital
Organization: Versailles Hospital (Other)
Other Study IDs: P24/08_ASCADA; 2024-A01041-46 (Other: ID RBC)
Record Dates: First submitted 2025-08-10; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-03

CONDITIONS: Coronary Artery Dilatations and Aneursyms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- aneurysmal or ectatic lesions of the coronary arteries: This is a non-interventional, observational, single-centre study conducted at the Centre Hospitalier de Versailles from 2013 to 2023, based on the department's coronary angiography registry. The study included adult patients, both living and deceased, who were hospitalised in the cardiology department and underwent coronary angiography between 1 January 2013 and 31 December 2023, which showed the presence of aneurysms or ectatic atheroma with bi- or tri-vessel coronary involvement.
  Interventions: Other: Anticoagulant Treatment

INTERVENTIONS:
Other: Anticoagulant Treatment — Follow-up of patients with coronary aneurysms and treatments introduced (anticoagulants and/or antiplatelet agents) to monitor the onset of ischaemic or haemorrhagic complications between 2013 and 2023.
  Other Names: Antiplatelet therapy

SUMMARY:
Objectives: The discovery of aneurysmal or ectatic lesions of the coronary arteries during coronary angiography or coronary CT angiography poses a triple challenge in terms of aetiology, treatment and prognosis. The aim of this study, based on coronary angiograms performed over a 10-year period at the Centre Hospitalier de Versailles, was to determine which antithrombotic treatment was routinely prescribed to patients with ACC or AEC, the evolution of this long-term treatment, and to analyse the association between the presence/absence of anticoagulant treatment and the rates of ischaemic cardiovascular events and haemorrhagic complications.

Materials and methods: This is a non-interventional, observational, single-centre study conducted at the Versailles Hospital Centre from 2013 to 2023, based on the department's coronary angiography registry. The study included adult patients, living or deceased, hospitalised in the cardiology department who underwent coronary angiography between 1 January 2013 and 31 December 2023, which showed the presence of aneurysms or ectatic atheroma with bi- or tri-vessel coronary involvement.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 years old
* Patient living or deceased
* Patient with aneurysmal or ectatic coronary artery disease with bi- or tri-truncular involvement at coronary angiography.

Exclusion Criteria:

* Patient < 18 years old
* Monotruncal aneurysmal or ectatic disease
* Absence of coronary aneurysm / ectasia
* Patient's opposition to participation in research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A patient with aneurysmal or ectatic coronary disease with bi- or tri-truncular involvement on coronary angiography.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2024-09-06 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2024-09-11 (Actual)

PRIMARY OUTCOMES:
The nature of the antithrombotic treatment prescribed between the initial hospital discharge and the follow-up date | Treatment on discharge from hospital and follow-up treatment beween 2013 and 2023
  The nature of the antithrombotic treatment prescribed between the initial hospital discharge and the follow-up date (anti-platelet agents alone, single or dual therapy, anticoagulant alone, anti-platelet agent-anticoagulant combinations).
The nature of antithrombotic treatments | Discharge from hospital (day 1)
  The nature of antithrombotic treatments

SECONDARY OUTCOMES:
The occurrence of ischaemic cardiovascular events (cardiovascular death, myocardial infarction, unscheduled coronary revascularisation) | The follow-up period between 2013 and 2023
  The occurrence of ischaemic cardiovascular events (cardiovascular death, myocardial infarction, unscheduled coronary revascularisation)
The occurrence of haemorrhagic events of any kind | The follow-up period between 2013 and 2025
  The occurrence of haemorrhagic events of any kind

CONTACTS AND LOCATIONS:
Overall Officials: Franck ASSAYAG, Principal Investigator — Versailles Hospital
Locations (1):
- Centre Hospitalier de Versailles, Le Chesnay, France